CLINICAL TRIAL: NCT02534181
Title: Refeeding Syndrome in Cancer Patients Admitted to Adult Intensive Care Unit
Brief Title: Refeeding Syndrome in Cancer Patients
Acronym: RESCUE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Logistical issues
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Eduardo Atsushi Osawa, ICU Consultant Physician, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1.015.415
Record Dates: First submitted 2015-08-23; First posted 2015-08-27 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Refeeding Syndrome; Cancer; Critical Illness
Keywords: Refeeding Syndrome; Cancer
MeSH Terms: conditions — Refeeding Syndrome; Neoplasms; Critical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Active Comparator): Patients will undergo a caloric management protocol:
  Days 1 and 2:
  1. Reduction of caloric intake to 5kcal/kg/day;
  2. Replacement of serum phosforus, potassium and magnesium;
  3. Administration of 100mg intravenous thiamine, vitamins and microelements.
  From day 3:
  1. If serum phosphorus < 2.5mg/dL, protocol will be followed according to day 2;
  2. If serum phosphorus > 2.5mg/dL, a gradual increase to target caloric intake will ensue.
  Interventions: Drug: Caloric Management Protocol
- Control group (No Intervention): 1. Nutritional management will be followed according to institutional protocol.
  2. Electrolyte replacement will be provided at the clinician's discretion.

INTERVENTIONS:
Drug: Caloric Management Protocol — Strategy based on reduction of nutritional intake and electrolyte replacement.
  Arms: Intervention group

SUMMARY:
The purpose of this study is to evaluate whether a nutritional strategy is effective in critically ill patients with cancer diagnosed with refeeding syndrome.

DETAILED DESCRIPTION:
Refeeding syndrome is a clinical entity triggered by the introduction of calories in chronically undernourished patients. A number of organs may be affected due to imbalance of fluids and electrolytes. In the intensive care setting, there are no formal guidelines to recommend the appropriate treatment of this condition. The aim of this study is to evaluate the implementation of a nutritional protocol to address cancer patients admitted to the ICU with refeeding syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Initiation of any type of nutrition (enteral, parenteral or glucose solution of at least 10% concentration) in the ICU in the last 48 hours;
* Reduction of serum phosphorus to a level below 2.5mg/dL with a drop above 0.5mg/dL compared to a previous measurement;
* Caloric intake greater than 500kcal in the last 24 hours;
* Central venous access for electrolyte replacement;
* Signature of the informed consent form.

Exclusion Criteria:

* Use of enteral or parenteral nutrition before ICU admission;
* Prediction of ICU discharge in the following 2 days;
* End-stage renal disease;
* Admission for diabetic ketoacidosis or hyperosmolar hyperglycemic state;
* Recent treatment of hyperphosphatemia;
* Parathyroidectomy surgery;
* Participation in another study;
* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Logistic Organ Dysfunction Score | 72 hours
  Score of the number and severity of organ failures during ICU stay

SECONDARY OUTCOMES:
ICU length of stay | 30 days
  Number of days in the ICU
Hospital length of stay | 30 days
  Number of days in hospital
Days in mechanical ventilation | 30 days
  Number of days in mechanical ventilation
Days in vasopressor therapy | 30 days
  Number of days using vasopressor therapy
Cardiovascular events | 30 days
  Incidence of acute ischemic event or acute heart failure
Delirium | 30 days
  Incidence of delirium according to CAM-ICU
Acute kidney injury | 30 days
  Incidence of acute kidney injury according to KDIGO
Mortality | 30 days
  Incidence of all-cause mortality
Renal Replacement Therapy | 30 days
  Number of days in renal replacement therapy
Acute ischemic stroke | 30 days
  Incidence of acute ischemic stroke
Seizures | 30 days
  Number of seizure episodes
Adverse events | 30 days
  Number of episodes of the following events: hypoglycemia, diarrhea, ileous, nausea and vomiting.

CONTACTS AND LOCATIONS:
Overall Officials: Ludhmila A Hajjar, MD, PhD, Study Chair — Director, Intensive Care Unit, Institute of Cancer of State of Sao Paulo; Eduardo A Osawa, MD, PhD, Study Director — Physician, Intensive Care Unit, Institute of Cancer of State of Sao Paulo; Ilana Roitman, Principal Investigator — Nutritionist, Intensive Care Unit, Institute of Cancer of State of Sao Paulo; Clarice H Park, MD, PhD, Principal Investigator — Physician, Intensive Care Unit, Institute of Cancer of State of Sao Paulo; Gisele Queiroz, MD, Principal Investigator — Physician, Intensive Care Unit, Institute of Cancer of State of Sao Paulo

REFERENCES:
- See also: Related Info — http://www.icesp.org.br